CLINICAL TRIAL: NCT02613884
Title: Safety, Efficacy, and Feasibility of High-dose Cholecalciferol in Pediatric Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 128487
Record Dates: First submitted 2015-11-20; First posted 2015-11-25 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Treatment (Experimental): All patients with a 25OHD level <30 ng/dL will be given 250,000 IU D3 (cholecalciferol) orally at one point in time and during CF clinic.
  Interventions: Drug: Treatment

INTERVENTIONS:
Drug: Treatment

SUMMARY:
Children with Cystic Fibrosis, ages greater than and equal to 36 months of age and less than or equal to 18 years of age, with a 25OHD level less than 30 ng/dL will be asked to participate in this study. Upon consent, they will be given oral cholecalciferol supplementation of 250,000 IU during their next CF clinic visit. The safety will be assessed by measuring a serum calcium level within 1 week of supplementation. Efficacy will be assessed using repeated 25OHD levels throughout the course of 12 months. Feasibility will be assessed with the previous two measures as well as a brief questionnaire administered via telephone within 1 week of supplementation.

DETAILED DESCRIPTION:
Children and adults with Cystic Fibrosis (CF) are at risk of developing a vitamin D deficiency or insufficiency, defined as a 2,25-hydroxyvitamin D (25OHD) serum blood level <30 ng/dL. Greater than 85% of people with CF have pancreatic insufficiency, which contributes to poor absorption of fat soluble vitamins in addition to dietary fat. A 25OHD level greater than 30 ng/dL has been described as providing potential improvements to markers of inflammation in adults with CF and is known to improve bone mineral density and prevent bone fractures in all populations, including CF. This study will assess the safety of a one-time high dose of cholecalciferol or vitamin D3 along with the efficacy and feasibility.

Children between the ages of 3 years and 18 years (inclusive), with a 25OHD level <30 ng/dL will be provided with a vitamin D3 supplement of 250,000 international units (IU) observed in our CF clinic. We hypothesize that this one-time, oral, high dose of vitamin D3 will safely and effectively raise the 25OHD level to above 30 ng/dL.

Safety will be monitored with serum calcium levels 1 week following the dosage, since 25OHD has a half-life of 2-3 weeks and this serum calcium level measurement time-point would be in or near the middle of this range. Feasibility will be measured using a 5-question phone survey 1 week following the dosage (see appendix A - attached). Efficacy will be measured by the 25OHD level itself; if 25OHD levels are found to be between 30-100 ng/dL over the course of the study, the dose will have demonstrated effective in achieving the study's goal.

The purpose of this study is to show that 25OHD levels can be safely corrected with a one-time dose of vitamin D3 that can be safely and feasibly provided in the outpatient setting to children with CF.

ELIGIBILITY:
Inclusion Criteria:

* Children with Cystic Fibrosis >36 months of age
* Serum/blood 25OHD level < 30 ng/dL
* Ability to provide valid informed consent to be a part of the study

Exclusion Criteria:

* Any history of kidney disease, kidney stones or on dialysis
* Any history of hypercalcemia
* Any history of hypercalciuria
* Pregnancy at time of enrollment
* Any history of parathyroid disorders
* Inability to swallow pills by mouth

Ages: 36 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2016-11; Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna Green, MD, Principal Investigator — Johns Hopkins All Children's Hospital
Locations (1):
- Johns Hopkins All Children's Hospital, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pediatric patients with Cystic fibrosis (CF) and greater than or equal to 36 months of age with a serum/blood 25OHD level < 30 ng/mL were recruited to participate in the study.
Groups:
- Treatment With High-Dose D3: All patients with a 25OHD level <30 ng/dL will be given 250,000 IU D3 (cholecalciferol) orally at one point in time and during CF clinic.
Period: Overall Study
Arm/Group | Treatment With High-Dose D3
Started | 26
Safety Endpoint 1 (Serum Calcium Level 1-week after dose) | 26
Feasibility Questionnaire (Phone survey) | 26
Safety Endpoint 2 (Serum Calcium Level at 3-month after dose) | 26
Efficacy Endpoint 1 (25OHD level at 3 Months) | 25
Efficacy Timepoint 2 (25OHD3 level at 6 months) | 25
Efficacy Timepoint 3 (25OHD3 level at 12 months) | 24
Completed | 24
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment: All patients with a 25OHD level <30 ng/dL & given 250,000 IU D3 (cholecalciferol).
Arm/Group | Treatment
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.46 (3.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 26
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
25-hydroxycholecalciferol (25OHD) level [Mean (Standard Deviation); unit: ng/mL] — The normal range for 25OHD is greater than or equal to 30 ng/mL.
  ng/mL | 22.69 (4.75)
Pancreatic Sufficient [Count of Participants; unit: Participants] — Pancreatic sufficiency is defined as a patient having enough exocrine pancreatic function to allow normal digestion without pancreatic enzyme supplementation.
  Participants
    Yes | 3
    No | 23
Taking additional vitamin D at enrollment [Count of Participants; unit: Participants]
  Yes | 18
  No | 8
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 20.09 (3.25)
BMI Percentile [Mean (Standard Deviation); unit: percentile] | 56.22 (24.21)

OUTCOME MEASURES:

1. Primary Outcome: Safety of a Single High-dose of Oral Cholecalciferol to Treat a Vitamin D Deficiency in Children With Cystic Fibrosis
Description: The safety of a single high-dose of oral cholecalciferol will be assessed using a serum calcium measurement after administration of treatment. Instances of hypercalcemia will be assessed at 1 week and at 3 months post-treatment. The treatment will be considered to be safe if the serum calcium level does not exceed 14 mg/dL.
Time Frame: 1 week, 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment With High-Dose D3
Number analyzed (Participants) | 26
mg/dL
  Serum Calcium 1-week | 9.57 (0.32)
  Serum Calcium 3-month | 9.47 (0.41)

2. Secondary Outcome: Efficacy of a Single High-dose of Oral Cholecalciferol in Treating a Vitamin D Insufficiency/Deficiency in Children With Cystic Fibrosis
Description: The efficacy of this treatment will be assessed by the 25OHD level measured after treatment at 3 months, 6 months, and 12 months. The treatment will be considered to be efficacious if the 25OHD level is greater than or equal to 30 ng/dL.
Time Frame: 3 months, 6 months and 12 months
Population: 26 participants were enrolled and given the treatment (250,000 IU D3) and assessed for the primary outcome measure. At the 3-month outcome measure, one participant had passed away, so 25 participants were included in the analysis. At the 12-month outcome measure, one additional participant was lost to follow-up, so 24 participants were included for analysis.
Measure: Mean (Inter-Quartile Range); unit: ng/dL
Arm/Group | Treatment
Number analyzed (Participants) | 25
ng/dL
  25OHD level at 3 months | 26 [24 to 31]
  25OHD level at 6 months | 30 [24 to 32]
  25OHD level at 12 months: number analyzed (Participants) | 24
  25OHD level at 12 months | 27 [22.5 to 30.2]

3. Secondary Outcome: Feasibility of Taking a 1-time High-dose of Cholecalciferol as Assessed by a 5-item Questionnaire
Description: CF patients with a 25OHD level <30 ng/dL who were given 250,000 IU D3. Feasibility will be measured using a 5-item Yes/No questionnaire where item 1 contains 5 sub-item yes/no questions which all relate to the experience of gastrointestinal symptoms. This was administered via telephone 1-week after administration of the treatment.
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With High-Dose D3
Number analyzed (Participants) | 26
Participants
  Increased amount of nausea: No | 24
  Increased amount of nausea: Yes | 2
  Increased frequency of emesis (vomiting): No | 26
  Increased frequency of emesis (vomiting): Yes | 0
  Increased amount of diarrhea?: No | 23
  Increased amount of diarrhea?: Yes | 3
  Any constipation?: No | 25
  Any constipation?: Yes | 1
  Increased gas production, such as burping or passing gas?: No | 24
  Increased gas production, such as burping or passing gas?: Yes | 2
  Increased amount of abdominal pain/stomach aches?: No | 23
  Increased amount of abdominal pain/stomach aches?: Yes | 3
  Incred in heart burn or reflux?: No | 24
  Incred in heart burn or reflux?: Yes | 2
  Easy to take?: No | 0
  Easy to take?: Yes | 26
  Something you would do next year if you had another low vitamin D level?: No | 0
  Something you would do next year if you had another low vitamin D level?: Yes | 26
  Prefer taking a one-time dose of vitamin D instead of a daily vitamin D?: No | 0
  Prefer taking a one-time dose of vitamin D instead of a daily vitamin D?: Yes | 26

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 1/26
Serious Adverse Events (participants affected / at risk) | 4/26
Other Adverse Events (participants affected / at risk) | 15/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=26)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Decreased lung function and weight loss (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchopneumonia exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=26)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Stomach ache (Gastrointestinal disorders) | 3 (3)
Increased burping (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Heart burn/Reflux (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxemia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elevated phosphorus level (General disorders) | 4 (4)
Elevated PTH (General disorders) | 1 (1)
Elevated calcium level (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT02613884/Prot_SAP_000.pdf